CLINICAL TRIAL: NCT00851695
Title: Vitamin D in Obstructive Lung Diseases
Brief Title: Examining the Role of Vitamin D in Asthma and Chronic Obstructive Pulmonary Disease (COPD)
Status: Completed | Type: Observational
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Augusto A. Litonjua, Assistant Professor, Brigham and Women's Hospital
Other Study IDs: 1399; R21HL089842-01 (NIH)
Record Dates: First submitted 2009-02-20; First posted 2009-02-26 (Estimated); Last update posted 2012-08-13 (Estimated); Status verified 2012-08

CONDITIONS: Asthma; Pulmonary Disease; Chronic Obstructive
Keywords: Lung Function Decline; Lung Function; Allergy; COPD; Vitamin D
MeSH Terms: conditions — Asthma; Lung Diseases; Hypersensitivity; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Serum samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Asthma: All 1024 participants of the Childhood Asthma Management Program, who provided blood samples.
- Asthma in Hispanics: All 616 subjects in the Genetic Epidemiology of Asthma in Costa Rica who have serum.
- Lung function and lung function decline: 626 subjects from the Normative Aging Study who have serum and lung function.

SUMMARY:
Asthma and chronic obstructive pulmonary disease (COPD) are diseases that affect a person's ability to breathe normally. People who do not receive enough vitamin D may have a higher risk of developing asthma or COPD. This study will examine previously collected blood samples of participants in three studies to determine whether people with low vitamin D levels have an increased risk of severe asthma or COPD.

DETAILED DESCRIPTION:
Asthma and COPD are among the leading causes of illness in children and adults, respectively. Asthma is the most common long-term disease among children in the developed world, and approximately 16 million people in the United States have COPD, which is now the fourth most common cause of death in this country. Vitamin D, both a nutrient and a hormone, can be taken in through diet and exposure to sunlight. Many children and adults have a vitamin D deficiency and there is concern that current recommended intake levels may be inadequate. A vitamin D deficiency can cause immune system dysfunction and may increase the risk of developing immune-mediated disorders, such as multiple sclerosis, inflammatory bowel disease, rheumatoid arthritis, and various cancers. Because of its role in immune development and function, a vitamin D deficiency may also be related to the development of severe asthma in children and to greater lung function decline in adults, leading to COPD. Preliminary research shows that people with asthma who take vitamin D have an enhanced response to corticosteroids, a common medication used to treat asthma. This finding suggests that vitamin D could possibly be used to improve asthma treatment. The purpose of this study is to measure vitamin D levels in participants of three previous studies and determine whether lower vitamin D levels are related to the development of severe asthma or COPD.

This study will examine previously collected blood samples from participants in three studies. There will be no study visits specifically for this study. The three studies include the following:

* Childhood Asthma Management Program, which is a study that examined the use of inhaled corticosteroids, nedocromil, and placebo in children with mild-to-moderate asthma
* Genetic Epidemiology of Asthma in Costa Rica, which is an ongoing study that is identifying genetic predictors of asthma in Costa Rican families with asthma
* Normative Aging Study, which is a study of aging that is being conducted in men living in Boston

ELIGIBILITY:
Inclusion Criteria:

* Participated in the Childhood Asthma Management Program, the Genetic Epidemiology of Asthma in Costa Rica study, or the Normative Aging Study

Ages: 5 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: For the Childhood Asthma Management Program, the study population was children with mild to moderate asthma, 5 to 12 years of age, living across the United States. For the Genetic Epidemiology of Asthma in Costa Rica study, the study population was children with asthma, 5 to 12 years of age, living in Costa Rica. For the Normative Aging Study, the study population was a community sample of men living in the Boston area.
Sampling Method: Non-Probability Sample
Enrollment: 2266 (Actual)
Dates: Start 2007-07; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Asthma exacerbation | Measured at Year 4 in the original study
Lung function decline | Measured at Year 15 in the original study

SECONDARY OUTCOMES:
Allergy markers | Measured at Year 4 in the original study

CONTACTS AND LOCATIONS:
Overall Officials: Augusto A. Litonjua, MD, MPH, Principal Investigator — Brigham and Women's Hospital